CLINICAL TRIAL: NCT03786809
Title: Vascular Effect of CIMICIFUGA RACEMOSA Versus Placebo Evaluated by Flow Mediated Dilatation of Brachial Artery (CRDILA)
Brief Title: Vascular Effect of CIMICIFUGA RACEMOSA
Acronym: CRDILA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Selmo Geber, Professor, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ETIC - CR-0417.0.203.000-09
Record Dates: First submitted 2018-12-21; First posted 2018-12-26 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Postmenopausal Symptoms
Keywords: postmenopause; vascular effects; CIMICIFUGA RACEMOSA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Women will use Cimifuga Racemosa for 28 days and will be submitted to measurement of the diameter of the brachial artery before and after treatment
  Interventions: Drug: Cimifuga Racemosa
- Placebo (Placebo Comparator): Women will use Placebo for 28 days and will be submitted to measurement of the diameter of the brachial artery before and after treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cimifuga Racemosa — Experimental group will use 160mg of Cimifuga Racemosa for 28 days
  Other Names: Clifemin; Acteia
  Arms: Experimental
Drug: Placebo — patients of the placebo group will use placebo once a day for 28 days
  Arms: Placebo

SUMMARY:
Postmenopausal women with vascular symptoms will use Cimifuga Racemosa or Placebo and the effects will be evaluated using Flow-Mediated Dilatation of the brachial artery.

DETAILED DESCRIPTION:
The interruption of the secretion of ovarian steroids after menopause, determines a change in the vascular pattern in several levels. Thus, several vascular effects might interfere with women's health. The use of hormone replacement therapy has contributed to the improvement in these effects. In previous studies, the investigators observed the effects of hormonal replacement therapy in improving such effects in postmenopausal women. The aim of the present study is to evaluate the effects of CIMICIFUGA RACEMOSA on the Flow-Mediated Dilatation of the brachial artery.

ELIGIBILITY:
Inclusion Criteria:

* Women with postmenopausal vascular symptoms
* Women without menstrual cycles within the last 12 months and follicle stimulating hormone (FSH) > 30 International Units(IU)/Litre
* Women that were not using drugs with potential vascular effect within the last 1 year
* Women that were not using hormone replacement therapy within the last 1 year

Exclusion Criteria:

* Smoking
* Blood Pressure > 160/90 mm Hg.
* Breast and or endometrial cancer
* History of acute myocardial infarction
* Diabetes
* Vaginal bleeding of any origin
* Hepatic disease
* Thrombophlebitis or thromboembolic disorders

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — only postmenopausal women will be included
Enrollment: 60 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Measurement of the brachial artery using flow-mediated dilation of post menopausal women, before and after use of Cimifuga Racemosa | 28 days
  We will evaluate the vascular effect of Cimifuga Racemosa on the brachial artery. The diameter of the artery will be measured before and one month after use of Cimifuga Racemosa and, in both situations, before and after the use of a cuff in the forearm. Measurement will be in millimeters.

SECONDARY OUTCOMES:
Frequency of symptoms and side effects | 28 days
  Patients symptoms before and after the use of Cimifuga Racemosa

CONTACTS AND LOCATIONS:
Overall Officials: Selmo Geber, MD PhD, Principal Investigator — Universidde Federal de Minas Gerais
Locations (1):
- Hospital das Clinicas - Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais, Brazil